CLINICAL TRIAL: NCT03364166
Title: Evaluation of Local Control in Buccinator Muscle Excision With the Skin Versus Buccinator Muscle Excision Without the Skin in Buccal Squamous Cell Carcinoma: A Randomized Clinical Trial.
Brief Title: Recurrence in Buccinator Muscle Excision With the Skin Versus Without the Skin in Buccal Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Yuseef, principle investigator, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: NCT
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
Keywords: buccal squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- buccinator muscle excision with skin (Active Comparator): surgical excision of the buccinator muscle with the skin in buccal squamous cell carcinoma and neck dissection also done
  Interventions: Procedure: surgical excision
- buccinator muscle excision without skin (Active Comparator): surgical excision the buccinator muscle without the skin in buccal squamous cell carcinoma and neck dissection also done.
  Interventions: Procedure: surgical excision

INTERVENTIONS:
Procedure: surgical excision — * Under general anaesthesia, the buccal squamous cell carcinoma which invaded the buccinator muscle will be excised with the skin of the cheek. This will be done by a safety margins in the soft tissue and the mandible may be resected according to the plan and the invasion of the tumour.
  * A neck dissection will be done in all cases of negative or positive neck lymph node.
  * Reconstruction of the soft tissue will be done immediately by a major pectorals flap with the skin, also bony reconstruction may be done by a reconstructed plate at the time of surgery then the patients will be prepared for bone graft in another surgery.

SUMMARY:
Evaluation of local control in buccinator muscle excision with the skin versus buccinator muscle excision without the skin in buccal squamous cell carcinoma: A randomized clinical trial.

DETAILED DESCRIPTION:
Preoperative Multi Slice CT scan or MRI carried out for evaluation the lymph node of the neck. Also, ultrasound carried out for measuring the depth of invasion of the tumour in the cheek (The invasion in the buccinator muscle).

* Under general anaesthesia, the buccal squamous cell carcinoma which invaded the buccinator muscle will be excised with the skin of the cheek. This will be done by a safety margins in the soft tissue and the mandible may be resected according to the plan and the invasion of the tumour.
* A neck dissection will be done in all cases of negative or positive neck lymph node.
* Reconstruction of the soft tissue will be done immediately by a major pectorals flap with the skin, also bony reconstruction may be done by a reconstructed plate at the time of surgery then the patients will be prepared for bone graft in another surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from buccal squamous cell carcinoma.
* Patients should be free from any systemic disease that may affect normal healing, and predictable outcome.
* Both sexes and all ages will be included in the study.
* Cooperative patients, who accept the procedure and return for follow up , examination and evaluation.

Exclusion Criteria:

* Patients with any systemic disease that may affect normal healing.9,10
* Patients who physically and psychologically not able to tolerate the procedures.
* Patients may discontinue the follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
local control | up to 1 year
  (recurrence rate)

CONTACTS AND LOCATIONS:
Overall Officials: ragia mounir, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided